CLINICAL TRIAL: NCT03197337
Title: Is Localized Provoked Vulvodynia Caused by Laxity of the Utero-Sacral Ligaments?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Prof. Jacob Bornstein, Chairman, Department of Obstetrics & Gynecology, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 004317NHR
Record Dates: First submitted 2017-06-22; First posted 2017-06-23 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Vulvodynia; Referred Pain
Keywords: Vulvodynia; Localized Provoked Vulvodynia (LPV); Referred pain; Utero-Sacral ligaments laxity
MeSH Terms: conditions — Vulvodynia; Pain, Referred

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants will not be informed prior to the experiment if they will first undergo the control manipulation or the study manipulation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control manipulation first (Experimental): Patients in this group will first undergo the control manipulation while the study manipulation will follow.
  Interventions: Procedure: Pressure-test
- Study manipulation First (Experimental): Patients in this group will first undergo the study manipulation while the control manipulation will follow.
  Interventions: Procedure: Pressure-test

INTERVENTIONS:
Procedure: Pressure-test — Pressure will be applied to the posterior fornix using a speculum.

SUMMARY:
Small-scale experiments conducted by our group have led to the hypothesis that Localized Provoked Vulvodynia (LPV) may be due to laxity of the Utero-Sacral ligaments (USL). According to this hypothesis, the pain experienced by women with LPV is due to the USL's inability to provide appropriate support for the pudendal nerve.

In order to test this hypothesis we will conduct a single-blind randomized control trial in which patients with LPV will undergo a pressure-test - pressure will be temporarily applied to the posterior fornix using a large-sized applicator, thus strengthening the USL and adding support to the pudendal nerve. While the pressure is being applied, the cotton-swab test will be performed (palpating vulvar and vestibular sites using a cotton-swab), and each patient will rate the elicited pain on a scale of 1 to 10 (1 - not painful, 10 - worst pain imaginable).

The results for each patient will be compared to their baseline level of pain (which will be recorded in the beginning of the experiment) and to the level of pain they report while inserting a speculum but not applying any pressure.

DETAILED DESCRIPTION:
Patients with LPV who sign an informed consent form will first undergo the cotton-swab test during which they will rate the pain elicited on a scale of 1 to 10. This score will be used as the patient's baseline level of pain for data analysis later. Then, each patient will be randomized into one of two groups: One group which will first undergo the control manipulation and then the study manipulation, or the second group in which the study manipulation will precede the control manipulation. This is done to neutralize a possible effect of the order of the manipulations on the trial's results when the data will be analyzed.

The control manipulation: Inserting a speculum into the vagina without applying pressure.

The study manipulation: First inserting a speculum, then inserting through it a large-sized applicator reaching the posterior fornix, then retrieving the speculum while keeping the applicator in place, and then applying significant pressure to the posterior fornix.

During each of the manipulations, the cotton-swab test will be performed again, and each patient will be asked to rate the level of pain elicited by the test. All data will be recorded, and we will later analyze if there was a significant difference between the pain elicited by the cotton-swab test during the study manipulation compared with the control manipulation, or compared with the baseline test.

ELIGIBILITY:
Inclusion Criteria:

* Women who suffer from LPV that are otherwise healthy.
* Symptoms severity in each patient is either moderate (able to engage in sexual intercourse despite suffering immense pain) or severe (unable to engage in sexual intercourse due to unbearable pain).
* Patients who have signed an informed consent form.

Exclusion Criteria:

* Women who suffer from Generalized Vulvodynia.
* Women who previously received other treatments for LPV, including but not limited to surgery, neuropathic treatment and/or physiotherapy.
* Women with uterine prolapse.
* Women who present with genito-urinary infection/inflammation at the day of the trial, or have healed from such a condition less then 14 days prior to the day of the trial.
* Women who have previously participated in clinical trials under which they received treatment for Vulvodynia.
* Women with LPV whose symptoms severity is defined as light (able to engage in sexual intercourse while suffering light pain / discomfort).
* Women who are pregnant at the day of the trial.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-07-23 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Level of pain | Immediate result
  Patients will rate the level of pain elicited each time the cotton-swab test will be performed, using a 1-10 scale (1 - not painful, 10 - worst pain imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bornstein, Prof, Principal Investigator — Chair, Obstetrics and Gynecology department
Locations (1):
- Department of Obstetrics and Gynecology, Nahariya, Israel

REFERENCES:
- [Background] Petros P, Bornstein J. Re: vulvar vestibulitis may be a referred pain arising from laxity in the uterosacral ligaments: a hypothesis based on three prospective case reports. Aust N Z J Obstet Gynaecol. 2004 Oct;44(5):484-5. doi: 10.1111/j.1479-828X.2004.00297.x. No abstract available. PMID 15387884
- [Background] Bornstein J, Zarfati D, Petros P. Re: Causation of vulvar vestibulitis. Aust N Z J Obstet Gynaecol. 2005 Dec;45(6):538-9. doi: 10.1111/j.1479-828X.2005.00499.x. No abstract available. PMID 16401228
- [Background] Friedrich EG Jr. Vulvar vestibulitis syndrome. J Reprod Med. 1987 Feb;32(2):110-4. PMID 3560069
- [Background] Bornstein J, Goldstein AT, Stockdale CK, Bergeron S, Pukall C, Zolnoun D, Coady D; consensus vulvar pain terminology committee of the International Society for the Study of Vulvovaginal Disease (ISSVD); International Society for the Study of Women's Sexual Health (ISSWSH); International Pelvic Pain Society (IPPS). 2015 ISSVD, ISSWSH, and IPPS Consensus Terminology and Classification of Persistent Vulvar Pain and Vulvodynia. J Sex Med. 2016 Apr;13(4):607-12. doi: 10.1016/j.jsxm.2016.02.167. Epub 2016 Mar 25. PMID 27045260